CLINICAL TRIAL: NCT04447807
Title: Rehabilitating Social Cognition: A Randomized Control Study Using Metacognitive Training in a Group Format With Bipolar Disorder Patients.
Brief Title: Metacognitive Training With Bipolar Disorder Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Beny Lafer, Associate Professor of the Department of Psychiatry (IPq), University of São Paulo Medical School, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4040551; 3148742040000068 (Other: CAAE)
Record Dates: First submitted 2020-06-08; First posted 2020-06-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Theory of Mind; Social Cognition; Metacognitive Training; Cognitive Rehabilitation; Cognitive Impairment
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients eligible for this study will be randomized into two groups: Metacognitive Training Intervention (9 weeks) or Treatment as Usual (9 weeks).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Metacognitive Training Intervention (Experimental): Participants of this group will undergo Metacognitive Training (MCT) in group format for the duration of 9 weeks. The intervention will be held once a week, with an estimated duration of 1-2 hours. The MCT intervention focuses on rehabilitating Social Cognition and teaching skills of interpersonal relations, as well as functional remediation aspects.
  We estimate a total of 26 participants in this group.
  Interventions: Behavioral: Metacognitive Training
- Group B: Treatment as Usual (Experimental): Participants of this group will continue to receive medical attention in the Bipolar Disorder Program -PROMAN- part of the University of São Paulo Medical School, although they will not be part taking in any group rehabilitation format We estimate a total of 26 participants in this group.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Metacognitive Training — MCT is a structured, interactive approach that addresses cognitive biases, social cognition, and self-esteem. This study will conducted this intervention using group format, on a weekly basis, with duration of 9 weeks total.
  Other Names: MCT
  Arms: Group A: Metacognitive Training Intervention
Other: Treatment as Usual — Patients will continue to receive medical attention in the Bipolar Disorder Program -PROMAN- part of the University of São Paulo Medical School.
  Other Names: TAU
  Arms: Group B: Treatment as Usual

SUMMARY:
The guiding question of this project is to evaluate the effectiveness of MCT as a form of ToM rehabilitation in patients diagnosed with BD who have deficits in this domain of social cognition. To do this, the work aims to be divided into three stages: (i) Evaluation of functionality through the FAST instrument (FAST score greater than or equal to 12 = mild impairment), to determine a subgroup of patients with deficits in functionality and evaluation scales for Montgomery & Åsberg Depression Rating Scale (MADRS) and Young Mania Rating Scale (YMRS) to verify euthymia, (ii) once these inclusion aspects have been verified, a neuropsychological assessment of hot cognition variables will be carried out, (iii) finally, the sample will be randomly divided into two groups, where one group will receive structured MCT rehabilitation and the other will continue with standard pharmacological treatment (TAU).

DETAILED DESCRIPTION:
The present study is justified by the importance of understanding, both theoretically and practically, psychotherapeutic interventions aimed at rehabilitating social cognition (SC) and specifically Theory of Mind (ToM) in individuals diagnosed with bipolar disorder (BD). ToM is an essential component for social interaction and, therefore, impairment in this area leads to problems related to interpersonal functioning. The majority of group rehabilitation interventions proposed for BD have focused primarily on cold cognitive domains or, in some cases, have only reserved one to two meetings to address strategies that integrate SC. BD is a heterogeneous disorder in terms of sociocognitive impairments and, therefore, demands more specific interventions for each individual ("personalized medicine"). Thus, the proposed intervention corresponds to a specific focus on functional rehabilitation of social cognition, with a focus on ToM and Emotion Recognition, and has not yet been evaluated in this population through a randomized controlled trial. Therefore, MCT intervention may be promising as a psychotherapeutic intervention for patients who present deficits in ToM (evaluated through their functionality).

Objectives

General Objectives To assess the overall effectiveness of MCT-BD (Metacognitive Training for Bipolar Disorder) in enhancing social cognition (theory of mind and emotion recognition) among euthymic individuals with Bipolar Disorder (BD).

Specific Objectives

Primary Efficacy Objectives:

1. To test the effectiveness of MCT-BD in improving Theory of Mind (ToM) among euthymic individuals with BD.
2. To test the effectiveness of MCT-BD in improving Emotion Recognition (ER) among euthymic individuals with BD.

Exploratory Objectives:

1. To assess the improvements in overall psychosocial functioning and quality of life of participants receiving MCT-BD compared to those receiving treatment as usual (TAU).
2. To assess the impact neurocognitive variables of participants receiving MCT-BD compared to those receiving treatment as usual (TAU)
3. To examine the effects of the intervention on mood variables within the same group.

General Objectives To assess the overall effectiveness of MCT-BD (Metacognitive Training for Bipolar Disorder) in enhancing social cognition among euthymic individuals with Bipolar Disorder (BD).

To deepen our understanding of social cognition in BD and lay the groundwork for tailored interventions aimed at improving psychosocial outcomes in this population.

Specific Objectives

Primary Efficacy Objectives:

To test the effectiveness of MCT-BD in improving Theory of Mind (ToM) among euthymic individuals with BD.

To evaluate the impact of MCT-BD on Emotion Recognition (ER) in the same population.

To assess the improvements in overall psychosocial functioning of participants receiving MCT-BD compared to those receiving treatment as usual (TAU).

Exploratory Objectives:

To investigate the impact of MCT-BD on neurocognitive variables in euthymic individuals with BD.

To examine the effects of the intervention on mood variables within the same group.

Hypothesis

We hypothesized that participants receiving MCT-BD would demonstrate significant improvements in:

Theory of Mind (ToM) Emotion Recognition (ER) Overall Psychosocial Functioning

Material and Methods

All participants will be recruited from patients regularly enrolled and clinically followed up at the Bipolar Disorder Program - PROMAN - outpatient clinic at Hospital das Clínicas, Faculty of Medicine, University of São Paulo. Participants will have access to the Informed Consent Form (ICF) for this research, and only those who agree to participate will be included in the study. This study aims to evaluate the efficacy of the MCT intervention with a specific focus on ToM and ER. To this end, the methodological proposal is divided into two stages: 01) Neuropsychological Evaluation of Cognition, ToM, and Social Cognition, and 02) MCT Intervention versus TAU.

Randomization Individuals with Bipolar Disorder recruited for the research will be randomized to the MCT arm or TAU arm through the Pass 22 tool using a true random algorithm.

Procedures All patients who meet the described criteria and agree to participate in the study by signing the research consent form will be evaluated using the proposed neuropsychological battery. To proceed to the next stage of the project (intervention), only patients who have a deficit (represented by a score of 12 or more points) on the functionality scale (Rosa et al., 2007) will be randomly distributed (using the Pass 22 tool and a true random algorithm by a third party blinded to the research) between the experimental (MCT) and control (TAU) groups. Twenty-six patients in the experimental group will participate in 9 weekly sessions following the MCT intervention proposal developed for this study. This will be based on a protocol recently developed for patients with TB by Haffner and colleagues (Haffner et al., 2018) and adapted and translated by the author of this project, Luisa de Siqueira Rotenberg, with authorization and approval for necessary modifications by the original authors. The other twenty-six patients in the control group will receive standard treatment (TAU). All patients will also be accompanied by medical consultations at the Bipolar Disorder Program outpatient clinic (PROMAN, IPq-HCFMUSP), which will be scheduled according to medical evaluation. The amount of medication used and the number of medical consultations will not be limited in this study, with the aim of increasing the generalization of possible results to real clinical situations. However, these variables will be subsequently observed through medical records produced during these consultations. The neuropsychological assessment battery will be applied to all participants before the start of therapy groups and will be reapplied after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of Bipolar Disorder Type I and Type II following the DSM-V criteria, using the Mini International Neuropsychiatric Interview (MINI) (Sheehan et al., 1998).
2. Adults between the ages of 18 and 60.
3. Both sexes.
4. FAST score greater than or equal to 12 (= mild impairment).
5. Education: Completed Elementary School, as a minimum educational criterion.
6. Estimated IQ ≥ 80.
7. Being in euthymia, assessed through scores lower than 8 on the Young Mania Rating Scale (YMRS) and/or 12 on the Montgomery-Åsberg Depression Rating Scale (MADRS).
8. Agreement to participate in the study by signing the Informed Consent Form (TCLE).

Exclusion Criteria

1. Subjects with complaints of visual or auditory sensory impairment that would not allow for the administration of the tests.
2. Subjects with organic mental disorders.
3. Subjects with a history of alcohol or drug abuse in the last six months.
4. Treatment with electroconvulsive therapy in the last 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Theory of Mind | Baseline and Follow-up (10 weeks)
  After the intervention, the group that received the MCT intervention will present changes from baseline Theory of Mind (ToM) scores at 9 weeks, when compared to TAU group. ToM Scores is evaluated by using Reading the Mind in the Eyes Test (RMET). Reading the Mind in the Eyes Test (RMET) is evaluated by each correct response is awarded 1 point, resulting in a minimum score of 0 and a maximum score of 28. Incomplete responses are treated as incorrect, domain scores are scaled in a positive direction (i.e. higher scores denote higher theory of mind).
Emotion Recognition | Baseline and Follow-up (10 weeks)
  Emotion Recognition will be evaluated through the subtask of the CANTAB: Emotion Recognition Task.CANTAB Emotion Recognition Task is a computer-based cognitive assessment tool designed to measure an individual's ability to recognize emotions from facial expressions. The task presents a series of faces, each displaying a different emotional expression, and the participant is required to identify the emotion being displayed (such as happiness, sadness, anger, or fear) by selecting the appropriate label from a list of options.

SECONDARY OUTCOMES:
Functioning Outcome | Baseline and Follow-up (10 weeks)
  The functional assessment scale (FAST): FAST is a standardized rating scale that is used to assess the functional impairment of individuals with bipolar disorder. The scale is designed to assess the level of functional impairment across a range of domains including autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, and leisure time. The FAST is typically administered as an interview-based assessment, with the interviewer asking questions about the individual's ability to perform specific tasks and activities in each of these domains.
Neuropsychological outcome | Baseline and Follow-up (10 weeks)
  The CANTAB subtests were chosen to provide objective measures of cognitive performance across domains such as reaction time, working memory, sustained attention, and verbal memory.
Quality of Life outcome | Baseline and Follow-up (10 weeks)
  The brief version of the World Health Organization Quality of Life questionnaire (WHOQOL-BREF) was utilized to evaluate global well-being subjectively.
Mood outcome measures | Baseline and Follow-up (10 weeks)
  The severity of manic and hypomanic symptoms was assessed using the Young Mania Rating Scale (YMRS) which comprises 11 items designed to evaluate the intensity of these symptoms The Montgomery Asberg Rating Scale (MADRS) was used to assess the severity of depression symptoms in patients. It consists of a 10-item questionnaire that evaluates various aspects of depression, quantitatively measuring symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Beny Lafer, Study Director — Associate Professor of the Department of Psychiatry, USP
Locations (1):
- Institute of Psychiatry, Clinic Hospital University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No